CLINICAL TRIAL: NCT05844748
Title: The Effect of Training Using Motivational Interview Technique in Type 2 Diabetes Patients on Perceived Self-Efficacy, Level of Adaptation to Disease and Metabolic Parameters
Brief Title: Motivational Interviewing in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sultan Yurtsever, Specialist diabetes nurse, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SYURTSEVER
Record Dates: First submitted 2022-12-05; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Motivation
Keywords: Diabetes Mellitus; Self-efficacy; Adaptation to illness; Behavior change; Motivational interview
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Motivational Interviewing Technique
Masking Description: 39 participants are in the intervention group and 39 participants are in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diabetes education with motivational interview technique (Experimental): A face-to-face motivational interview session was applied to each participant in the experimental (intervention) group by the researcher once a week in the 1st month and once in 15 days in the 2nd month. The interviews were held in 6 sessions in total, and each interview was completed in approximately 45-60 minutes.
  Interventions: Other: diabetes education with motivational interview technique

INTERVENTIONS:
Other: diabetes education with motivational interview technique — Techniques such as developing empathy, developing disengagement, turning with resistance, supporting self-efficacy, avoiding advice, a simple decision, importance-trust scale, open-ended questions, reflection and segmentation in motivational interviews.
  Other Names: general method of diabetes education

SUMMARY:
This research was planned to examine the effects of diabetes education given by motivational interviews on adherence to the disease, perception of diabetes self-efficacy and metabolic parameters in diabetes patients. The research sample will consist of 78 individuals with type 2 diabetes (39 intervention group - 39 control group). Diabetes education will be given to the participants in the intervention (experimental) group of the research with the motivational interview method based on the Transtheoretic Model. The interviews will be completed at the end of 2 months, with a total of 6 sessions in the first month (4 sessions per month) and once every 15 days in the 2nd month (2 sessions per month). Participants in the control group will be given standard diabetes education. Participants in the intervention (experimental) and control groups will be asked to follow the habit of exercising regularly and blood sugar.

DETAILED DESCRIPTION:
To the participants in the intervention group of the research; Diabetes education will be given by using the motivational interview method, which is structured on the basis of the Transtheoretic Model. Data will be obtained by face-to-face interview method individually. Information will be obtained from the following forms as a pre-test for the participants in the initiative group:Patient Information Form [App. 1], Behavioral Change Stage Diagnosis Form in Patients with Type 2 Diabetes [App. 2], Diabetes Self-Efficacy Perception Scale [App. 3], Chronic Disease Adjustment Scale [App. 4]. Metabolic parameters of patients before the motivational interview Metabolic Results It will be recorded in the Follow-up Form (HbA1c, FCC, HDL cholesterol, LDL cholesterol, Triglyceride, Total Cholesterol, Height, Weight, BMI) [App. 5].Diabetes education will be given to the intervention (experimental) group using the motivational interview method consisting of 6 sessions. The interviews will be completed at the end of 2 months, with a total of 6 sessions in the first month (4 sessions per month) and once every 15 days in the 2nd month (2 sessions per month). The participants in the intervention group will be given a Blood Glucose Follow-up Chart [App. 6] at the first meeting, and they will be asked to bring the Blood Glucose Follow-up Chart with them at each meeting (6 times in total), by writing the follow-up result. After explaining the positive effect of exercise on blood glucose to the participants in the intervention group, the Walking Program Implementation Chart will be given. Participants will be asked to record the total number of steps per day, together with the date they walked, the number of steps taken during walking, and any complaints experienced, and bring them together in each motivational interview session (6 times in total).In the first interview, the researcher will provide and give the individual the Walking Program Implementation Chart, along with the pedometer that they will use to track the number of steps in their daily activities. In each motivational interview session, the individual's daily step counts will be checked. At the end of the first session, the participants in the intervention group will be given the "Educational Guide for Individuals with Diabetes" booklet, which will be prepared by the researcher. Participants in the intervention group will be informed by the researcher via reminder phone messages (SMS) once a week (6 times in total) to exercise regularly.As a post-test for the participants in the intervention group; Patient Information Form [App 8], Behavior Change Stage Diagnosis Form in Patients with Type 2 Diabetes [App. 2], Diabetes Self-Efficacy Perception Scale [App. 3], Chronic Disease Adjustment Scale [App. 4]. Diabetes education of the participants in the intervention group using motivational interview method Blood glucose and lipid profile will be monitored as metabolic parameters and recorded in the Metabolic Results Follow-up Form [App. 5] at the 3rd month after completion. The height and weight follow-up of the participants in the intervention group will be done again in the 3rd month after the end of the motivational interview sessions and recorded in the Metabolic Results Follow-up Form [App. 5] by the researcher.As a pre-test before starting the general diabetes education among the participants in the control group; Patient Information Form [App. 1], Behavioral Change Stage Diagnosis Form in Patients with Type 2 Diabetes [App. 2], Diabetes Self-Efficacy Scale [App. 3], Chronic Disease Adjustment Scale [App. 4] will be used.Metabolic Results (HbA1c, FCC, HDL, LDL, Triglyceride, Total Cholesterol, Height, Weight and BMI) Follow-up Form [App. 6], Individual general diabetes education lasting 30-60 minutes on average will be given to the participants in the control group. At the 3rd month after general diabetes education, participants in the control group will be asked to complete the posttests again (App. 2,3,4,8). The metabolic parameters of the participants in the control group will be monitored in the 3rd month and recorded by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 18 and under 65.
* Must be diagnosed with diabetes type 2 and treated for more than 6 months
* Must able to understand and speak Turkish.
* Must volunteer to participate in the research.

Exclusion Criteria:

* Being younger than 18 years of age
* Being at the age of 65 or older
* Reluctance to participate in the research.
* Type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The Effect of Training Given by Motivational Interview Technique on Self-Efficacy Perception, Level of Adjustment to Disease and Metabolic Parameters in Type 2 Diabetes Patients | 3 mounth
  After diabetes education given by motivational interviews It is expected that there will be an increase in the level of self-efficacy and compliance with the disease, and an improvement in metabolic parameters in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study, which was planned and carried out as a doctoral thesis, will be published scientifically after the completion of the research.
Supporting Information: CSR
Time Frame: 2024-2025
Access Criteria: This study will be shared with nurses giving care to diabetes patients and aims to benefit type 2 diabetes patients
URL: https://tez.yok.gov.tr/

REFERENCES:
- See also: Tip 2 Diyabet Tanılı Yetişkinlerde Motivasyonel Görüşmenin Etkisi: Sistematik Derleme * — https://dergipark.org.tr/en/download/article-file/752953
- See also: Tip 2 Diabetes Mellitus'ta Sağlık Davranış Değişiminde Transteoretik Model Temelli Motivasyonel Görüşme Tekniği — https://dergipark.org.tr/tr/download/article-file/115235